CLINICAL TRIAL: NCT05057325
Title: Post Operative Pain After Pulpectomy of Primary Molars With One Shap Rotation File Versus Wave One Reciprocating File
Brief Title: Post Operative Pain Assessment After Pulpectomy of Primary Molars With Two Different Rotary Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 605
Record Dates: First submitted 2021-08-30; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Pulp Necroses
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wave One Gold (Experimental): Receporcating single file used for preparation of root canals in primary molars
  Interventions: Other: Pulpectomy using single file system ( WaveOne Gold file)
- One shape (Experimental): Rotation single file used for preparation of root canals in primary molars
  Interventions: Other: Pulpectomy using single file system ( One Shape file)

INTERVENTIONS:
Other: Pulpectomy using single file system ( One Shape file) — Rotary file instrument for pulpectomy of primary molars ( One shape file)
  Arms: One shape
Other: Pulpectomy using single file system ( WaveOne Gold file) — Rotary file instrument for pulpectomy of primary molars ( WaveOne Gold file)
  Arms: Wave One Gold

SUMMARY:
Evaluation of post operative pain after pulpectomy procedures for primary molars with irreversible pulp damage and without periapical radulicency using two different systems (One shape file ( ratation movemont) and wave one gold file ( reciprocation movement)

ELIGIBILITY:
Inclusion Criteria:

* Age of more than 4 years
* Healthy children
* Primary molars with irreversible pulp damage

Exclusion Criteria:

* Presence of periapical radiolucency realtes to primary molar
* Uncooperative child

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 164 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 1 week
  Assessment of pain using 4 piont intensity scale
  1 means no pain, 2 means slight pain, 3 means moderate pain and for means sever pain at 6,12, 48,72 hours and 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt